CLINICAL TRIAL: NCT01582633
Title: Assessment of Dose-sparing of Pandemic A/California/7/2009 H1N1 Influenza Vaccine Administered Intradermally by Needle-free Disposable-syringe Jet Injector (DSJI)
Brief Title: Assessment of Needle-free Disposable-syringe Jet Injector (DSJI) ID Dose-sparing of Pandemic A H1N1 Influenza Vaccine
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: D'Antonio Consultants International, Inc. (Other); Sao Paulo, Secretaria de Estado da Saúde (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAPPesq 0015/2010
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Influenza
Keywords: vaccine; influenza; needle free jet injector; Intradermal; sparing dose
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.1 ml ID dose (Experimental): Dose of 0.1 ml ID trivalent 2012 influenza vaccine administered by disposable needle-free jet injector
  Interventions: Biological: 2012 trivalent influenza vaccine
- 0.2 ml ID dose (Experimental): Dose of 0.2 ml ID trivalent 2012 influenza vaccine administered by disposable needle-free jet injector
  Interventions: Biological: 2012 trivalent influenza vaccine
- 0.5 ml IM dose - needle-free (Experimental): Dose of 0.5 ml IM trivalent 2012 influenza vaccine administered by disposable needle-free jet injector
  Interventions: Biological: 2012 trivalent influenza vaccine
- 0.5 ml IM - needle and syringe (Active Comparator): Dose of 0.5 ml IM trivalent 2012 influenza vaccine administered by needle and syringe
  Interventions: Biological: 2012 trivalent influenza vaccine

INTERVENTIONS:
Biological: 2012 trivalent influenza vaccine — 2012 trivalent influenza vaccine:
  * influenza A/California/7/2009 (H1N1)
  * influenza A/Perth/16/2009 (H3N2)
  * influenza B/Brisbane/60/2008 Single dose.

SUMMARY:
This study will evaluate the immunological response and the safety profiles of seasonal, inactivated vaccine which contains in its composition the A/California/7/2009 H1N1 "pandemic" influenza virus, delivered via ID in reduced dose (0,1 mL) and (0,2 mL), and via IM in full dose (0,5 mL) delivered with needle-free, disposable-syringe jet injector, and control group with via IM in full dose (0,5 mL) delivered syringes and needles in subjects from 42 to 60 years old.

Reduced doses into the skin will be delivered by an investigational intradermal model of a licensed, needle-free, disposable-syringe jet injector (DSJI) system, LECTRAJET® M3 RA manufactured by D'Antonio Consultants International, Inc. DSJIs avoid the drawbacks and dangers of conventional needle-syringe injection. Delivery by DSJI into the skin is also rapid and simple and overcomes the difficulty and patient discomfort of the traditional Mantoux needle method for skin injection, as used for BCG vaccination and tuberculosis skin testing.

Participants will be assessed for local and systemic adverse events by clinical observation immediately after injection and then upon return on day 21 after each injection. In addition, investigators will call participants by telephone on days 2 and 7 days to collect information local and systemic side effects.

Serum will be collected on day 21 after each injection, and assayed for hemagglutination inhibition (HAI) using conventional methods performed by the Virology Lab of the Instituto de Medicina Tropical de São Paulo, blinded to the study arm allocations of each participant. Information about the adverse events would be collected on days 1, 3 and 7 after dose delivery. The investigators assessing adverse reactions will be blinded to the study arm to which each subject was allocated.

The primary endpoint of the study is to evaluate the vaccine's immunogenicity by HAI, each dose in accordance with international parameters which include: seroconversion or significant title increase (SCR), the frequencies by study arm of seroprotection defined as a post-vaccination titer of >40 (1/dil) (SPR), as well as the Geometric Mean Titers (GMTRs) of post-vaccination sera.

DETAILED DESCRIPTION:
This study will evaluate the immunological response and the safety profiles of seasonal, inactivated vaccine which contains in its composition the A/California/7/2009 H1N1 "pandemic" influenza virus, delivered via ID in reduced dose (0,1 mL) and (0,2 mL), and via IM in full dose (0,5 mL) delivered with needle-free, disposable-syringe jet injector, and control group with via IM in full dose (0,5 mL) delivered syringes and needles in subjects from 42 to 60 years old.

Reduced doses into the skin will be delivered by an investigational intradermal model of a licensed, needle-free, disposable-syringe jet injector (DSJI) system, LECTRAJET® M3 RA manufactured by D'Antonio Consultants International, Inc. ( East Syracuse, NY, USA) . DSJIs avoid the drawbacks and dangers of conventional needle-syringe injection. Delivery by DSJI into the skin is also rapid and simple and overcomes the difficulty and patient discomfort of the traditional Mantoux needle method for skin injection, as used for BCG vaccination and tuberculosis skin testing.

Participants will be assessed for local and systemic adverse events by clinical observation immediately after injection and then upon return on day 21 after each injection. In addition, investigators will call participants by telephone on days 2 and 7 days to collect information local and systemic side effects. Adverse events will be classified and analyzed according to case definitions established by the Brighton Collaboration Group.

Serum will be collected on day 21 after each injection, and assayed for hemagglutination inhibition (HAI) using conventional methods performed by the Virology Lab of the Instituto de Medicina Tropical de São Paulo, blinded to the study arm allocations of each participant. Information about the adverse events would be collected on days 1, 3 and 7 after dose delivery. The investigators assessing adverse reactions will be blinded to the study arm to which each subject was allocated.

The primary endpoint of the study is to evaluate the vaccine's immunogenicity by HAI, each dose in accordance with international parameters which include: seroconversion or significant title increase (SCR), the frequencies by study arm of seroprotection defined as a post-vaccination titer of >40 (1/dil) (SPR), as well as the Geometric Mean Titers (GMTRs) of post-vaccination sera.

Participants will be excluded if they have a prior history of influenza disease caused by A/California/7/2009 H1N1 or prior vaccination for same, among other exclusion and inclusion criteria to apply. Participants will be excluded retroactively from analysis if their pre-vaccination HAI assay discovers pre-existing seroprotective titers of >40 against pandemic virus, representing preexisting H1N1 exposure or vaccination

ELIGIBILITY:
Inclusion Criteria:

* Between 42 and up to 60 years of age.
* Available for follow up visits, at least at day 21.
* Written informed consent signed by the volunteer after reading and explanation.

Exclusion Criteria:

* Suspect or verified diagnosis of congenital or acquired immunodeficiency including AIDS.
* Suspect or verified diagnosis of malignant neoplasia, other than basocellular carcinoma.
* Volunteer ongoing treatment with high doses of systemic corticosteroids (equivalent to prednisone (2 mg/kg/d for more than two weeks) or on immunosuppressant therapy.
* Received or planning to receive a vaccine with live attenuated strain of virus within 30 days of the intended day(s) of study vaccination(s).
* Verified diagnosis of Influenza A/California/H1N1 or has already been immunized against (Influenza A/California/H1N1).
* Suspect or confirmed pregnancy (no need of pregnancy test, information on possible pregnancy is enough. These cases must be referred to routine vaccination).
* Suspect or verified diagnosis of hypersensitivity to any ingredient of the vaccine, to egg proteins or any component of the vaccine or life-threatening reactions after previous administration of any influenza vaccine.
* Any other circumstances that may potentially damage the minor or prevent procedures from being carried out according to evaluation of the research team.
* Volunteer shows signs or symptoms of an active intercurrent disease (e.g. fever, rash, etc.) that may interfere with the evaluation of adverse events following immunization at the research team's discretion.

Ages: 42 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | 21 days
  Assess whether the experimental and standard dosages/delivery routes (ID and IM) for each age group met all modified criteria for assessment of influenza vaccines 21 days after vaccination for soroconversion for A/California/7/2009 H1N1 influenza virus.

SECONDARY OUTCOMES:
Safety | 21 days
  Evaluate frequency and severity of local and systemic adverse events following immunization between investigational (reduced dose) and control (standard dose) adult groups up to 21 days after vaccination in accordance with the definitions of the Brighton Collaboration Group.
Seasonal influenza immunogenicity | 21 days
  Assess whether the experimental and standard dosages/delivery routes (ID and IM) for each age group met all modified criteria for assessment of influenza vaccines 21 days after vaccination for soroconversion for 2012 seasonal influenza viruses.

CONTACTS AND LOCATIONS:
Overall Officials: Glacus Brito, MD, Principal Investigator — Hosp das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo
Locations (1):
- Hosp das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil